CLINICAL TRIAL: NCT03041675
Title: Effects of Laser Acupuncture Therapy on Paralytic Ileus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMUH105-REC1-133
Record Dates: First submitted 2017-01-23; First posted 2017-02-03 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Paralytic Ileus
Keywords: Lacer Acupuncture; Paralytic ileus
MeSH Terms: conditions — Intestinal Pseudo-Obstruction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser Acupuncture group (Experimental): 47 participants receive 10 seconds of Laser Acupuncture(808nM/300mW) on acupoints RN6, RN4, and RN12. The whole duration of treatment is 3 times a week, for 8 weeks.
  Interventions: Device: Laser Acupuncture group
- Sham Laser Acupuncture group (Sham Comparator): The investigators apply the Laser Acupuncture pen (without pressing the laser button) on other 47 participants' acupoints RN6, RN4, and RN12. The whole duration of treatment is 3 times a week, for 8 weeks.
  Interventions: Device: Sham Laser Acupuncture group

INTERVENTIONS:
Device: Laser Acupuncture group — 47 participants receive 10 seconds of Laser Acupuncture(808nM/300mW) on acupoints RN6, RN4, and RN12. The whole duration of treatment is 3 times a week, for 8 weeks.
  Arms: Laser Acupuncture group
Device: Sham Laser Acupuncture group — The investigators apply the Laser Acupuncture pen (without pressing the Laser button) on other 47 participants' acupoints RN6, RN4, and RN12. The whole duration of treatment is 3 times a week, for 8 weeks.
  Arms: Sham Laser Acupuncture group

SUMMARY:
Ileus occurs from hypomotility of the gastrointestinal tract. Causes of Paralytic ileus include post-operation, stroke, and bed-ridden for a long time. Medicine treatment is less and less effective over time. Some study revealed that Moxibustion and Acupuncture are effective in Paralytic ileus. Investigators try to find other treatment except of medicine. Laser Acupuncture is a safe and non-invasive choice. This study is to evaluate effect of Laser Acupuncture on Paralytic ileus.

DETAILED DESCRIPTION:
This study's sample consisted of 94 adult participants who had Paralytic ileus. Patients experiencing skin disease or wounds, pregnancy, less than 20 years old, and who take Immunosuppressants drugs or Morphine, Mechanical obstruction were excluded. These 94 patients were randomly divided into two groups: a Laser Acupuncture group and a control group. At the beginning of study, check X-ray(KUB), collect serum Gastrin, Motilin, and Pancreatic polypeptide, and record bowel sound per minute, frequent of enema, average amount of stool per day. 47 patients received Laser Acupuncture therapy three times a week in acupoints RN6, RN4, and RN12. The whole duration of treatment is 8 weeks. The control group patients receive pseudo laser acupuncture. In the end of 4th and 8th week, check X-ray(KUB), collect serum Gastrin, Motilin, and Pancreatic polypeptide, and record bowel sound per minute, observe the daily record and then calculate frequent of enema and average amount of stool per day. After the end of treatment, the investigators keep follow up for 4 weeks. The outcome parameters include:

1. KUB,
2. the average amount of stool every day,
3. frequency of bowel sound,
4. frequency of enema, (Indication of enema: the amount of stool less than 200g within 3 days),
5. the change of serum Gastrin, Motilin, and Pancreatic polypeptide.

ELIGIBILITY:
Inclusion Criteria:

* Already sign test consent permit.
* More than 20-year-old.
* Doctors diagnosis as Paralysis ileus, and KUB report was improved as Paralysis ileus by Radiologists.

Exclusion Criteria:

* Pregnant.
* Patients taking immunosuppressive or morphine analgesics.
* Skin infections.
* Without test consent permit.
* mechanical ileus, mechanical obstruction.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2017-02-13 (Estimated); Primary Completion 2017-06-30 (Estimated); Study Completion 2017-08-31 (Estimated)

PRIMARY OUTCOMES:
the changing of diameter of colon (KUB) | the 4th, 8th, 12th week
  Definition of Ileus: Diameter of colon: >6cm. Check KUB on the 4th, 8th, 12th week. Calculate the biggest diameter of colon. Is diameter of colon decreasing in Laser Acupuncture group?

SECONDARY OUTCOMES:
the average amount of stool per day(g/Day) | the 4th, 8th, 12th week
  Is the average amount of stool per day elevating in laser group?

OTHER OUTCOMES:
bowel sound | the 4th, 8th, 12th week
  Record frequency of bowel sound. Is bowel sound increased after Laser Acupuncture
frequency of enema | the 4th, 8th, 12th week
  Is frequency of enema decreasing in laser group?(Indication of enema: the amount of
serum Gastrin (pmol/L) elevation | the 4th, 8th, 12th week
  Gastrin is secreted by G cell at stomach. It stimulates parietal cells of the stomach to secrete hydrochloric acid (HCl)/gastric acid. It also increases antral muscle mobility and promotes stomach contractions. Collect serum 3cc before study, and on the end of 4th, 8th, 12th week. Check serum Gastrin. Is serum Gastrin increased after Laser Acupuncture Therapy?
serum Motilin (pmol/L) elevation | the 4th, 8th, 12th week
  Motilin is secreted by endocrine M cells that are numerous in crypts of the small intestine, especially in the duodenum and jejunum. It's the most important factor in controlling the inter-digestive migrating contractions. Collect serum 3cc before study, and on the end of 4th, 8th, 12th week. Check serum Motilin. Is serum Motilin increased after Laser Acupuncture Therapy?
serum Pancreatic polypeptide (pmol/L) elevation | the 4th, 8th, 12th week
  Pancreatic polypeptide is released mainly from the pancreas. Pancreatic polypeptide has been shown to stimulate colonic muscle contraction. Collect serum 3cc before study, and on the end of 4th, 8th, 12th week. Check serum Pancreatic polypeptide. Is serum Pancreatic polypeptide increased after Laser Acupuncture Therapy?

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang JS, Lee SB, Park SY. The effect of SSP therapy on elderly nursing home residents' chronic constipation. J Phys Ther Sci. 2015 Dec;27(12):3887-9. doi: 10.1589/jpts.27.3887. Epub 2015 Dec 28. PMID 26834374
- [Background] Moriya R, Fujikawa T, Ito J, Shirakura T, Hirose H, Suzuki J, Fukuroda T, Macneil DJ, Kanatani A. Pancreatic polypeptide enhances colonic muscle contraction and fecal output through neuropeptide Y Y4 receptor in mice. Eur J Pharmacol. 2010 Feb 10;627(1-3):258-64. doi: 10.1016/j.ejphar.2009.09.057. Epub 2009 Oct 8. PMID 19818748
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/19818748